CLINICAL TRIAL: NCT03138746
Title: Insulin Sensitivity During Hyperbaric Oxygen Compared to Hyperbaric Air
Acronym: HOTAIR4
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Collaborators: Royal Adelaide Hospital (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, ARC Future Fellow, University of Adelaide
Other Study IDs: R20160801
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type II; Insulin Resistance
Keywords: hyperbaric oxygenation; insulin sensitivity; human; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HBO: On day 2, the participant will undergo a 2-hour hyperbaric exposure breathing 100% oxygen
  Interventions: Procedure: HBO
- Hyperbaric air: On day 2, the participant will undergo a 2-hour hyperbaric exposure breathing air
  Interventions: Procedure: Hyperbaric air

INTERVENTIONS:
Procedure: HBO — Compression in a hyperbaric chamber in air to 2 atmospheres absolute, then donning a "hood" supplying high flow oxygen for 90-minutes followed by a linear decompression back to 1 atmosphere over 30 minutes
  Groups: HBO
Procedure: Hyperbaric air — Compression in a hyperbaric chamber in air to 2 atmospheres absolute, then donning a "hood" supplying high flow air for 90-minutes followed by a linear decompression back to 1 atmosphere over 30 minutes
  Groups: Hyperbaric air

SUMMARY:
In a recent series of studies performed by our group, we have shown that exposure to hyperbaric oxygen (HBO) leads to an increase in insulin sensitivity in male subjects with type-2 diabetes (T2DM) and in obese and overweight men without diabetes. The aim of this study is to investigate the relationship between pressure and oxygen in producing this effect, specifically, is this effect measurable in hyperbaric air or is some higher pressure of oxygen required?

Aims:

1. To determine whether the insulin sensitising effect of HBO is apparent in hyperbaric air at the same pressure as HBO.
2. To examine mechanisms underpinning the increase in insulin sensitivity following HBO.

DETAILED DESCRIPTION:
The 40 participants will be randomly allocated to two groups, matched for BMI. All participants will attend the Hyperbaric Medicine Unit on 2 occasions and metabolic testing will be undertaken at the same time of the day. Day 1 will be for baseline assessment sitting outside the hyperbaric chamber. Day 2 will be two days after Day 1 in the same week during which participants will undergo a 2-hour session in the hyperbaric chamber with a "10:90:30" compression profile (compression of the chamber in air to 2 atmospheres absolute, then donning a "hood" supplying high flow gas for 90-minutes followed by a linear decompression back to 1 atmosphere absolute over 30-minutes). Half of the participants will breathe oxygen during this compression profile while the other half will breathe medical air.

An overnight fast (10-hours) will be required prior to each day with modification of their diabetic medication. This regimen will be monitored in consultation with a diabetes specialist (IC):

* If prescribed metformin, withhold the evening dose before each study day but give other usual evening oral drugs
* If taking evening insulin, reduce dose to 2/3 of usual dose the night before each study day
* Hold diabetes drugs (oral or injectable) on morning of study until conclusion of study and then administer with food. Take usual morning oral medication at this time and modified insulin dose (if prescribed insulin)
* Check BSL on arrival and departure each study day

Day 1. Baseline assessment. The participant will attend at 0900 for a hyperinsulinaemic euglycaemic clamp, which will be performed with the same protocol as used in our three previous clamp studies. Two intravenous cannulae are inserted into veins in contralateral forearms using local anaesthetic (lignocaine 1%). Baseline blood is taken for fasting glucose and insulin and a primed insulin infusion is started (80mU/m2/min) for 3½ hours. Blood samples (<2mls) are obtained at 5-10 minute intervals so that blood glucose can be maintained at 5.5 mmol/L with a variable infusion of 25% Dextrose and a trained individual will be present for the duration of the clamping procedure. Insulin sensitivity will be assessed by the steady state glucose infusion rate calculated over a stable 30-minute period of the clamp. Assessments will be made at two points during the 3½ hour clamp; at 2½-3 hours and 3-3½ hours. Immediately post-clamp, volunteers are given orange juice and high carbohydrate lunch, and the glucose infusion is maintained on halving scale for 5 minutes each for at least 20 minutes. Blood sugar levels are monitored every 10-15 minutes for 60 minutes. Total blood taken during the clamping procedure will be less than 100mls including baseline samples. The researchers have performed several hundred clamps.

Day 2. The participant will attend at 0900 for a second 3½-hour hyperinsulinaemic euglycaemic clamp, similar to Day1. The procedure for the two groups (HBO and hyperbaric air) will be identical, the only difference will be the breathing gas used during the 10:90:30 hyperbaric exposures. The breathing gas delivered to the participant (oxygen or air) will be supplied from masked "research" gas outlets, so the participant will be blinded as to which group they are in. The participant will enter the chamber after a 1-hour clamp stabilising period and assessment of the steady state glucose infusion rate will take place at similar times to Day1. This means that during the 2-hour hyperbaric exposure, the assessment periods will correspond to the 30-minute decompression at the end of the hyperbaric session and the first 30-minutes after exit from the hyperbaric chamber. Post clamp will be managed as during Day1.

Blood samples (20 ml) for inflammatory markers will be taken before and after procedures on both days. With blood taken during 2 clamps (less than 100mls each) and four 20 ml samples, total blood taken will be approximately 280 ml.

ELIGIBILITY:
Inclusion Criteria:

* Men with T2DM, n=40 (numbers are based on power analysis of previous studies)
* Normal to obese weight (BMI 25-40 kg/m2)
* Age > 40 (no specific upper age limit)
* All participants will attend the Hyperbaric Medicine Unit to be assessed by a hyperbaric physician (DW) to determine fitness to enter the hyperbaric chamber the standard clinical criteria of the Hyperbaric Medicine Unit will be used

Exclusion Criteria:

* use of prescribed or non-prescribed medications which may affect glucose homeostasis (eg steroids)
* uncontrolled asthma, current fever, upper respiratory infections
* individuals who regularly perform high intensity exercise (>2 week)
* current intake of > 140g alcohol/week
* current smokers of cigarettes/cigars/marijuana
* current intake of any illicit substance
* experience claustrophobia in confined spaces
* has donated blood within past 3-months
* has been involved in any other study within the past 3-months
* unable to comprehend study protocol
* any other contraindication to HBO (eg Eustachian tube dysfunction making middle ear inflation ineffective)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | Baseline to Day 2
  As measured by the glucose infusion rate during the steady-state phase of the hyperinsulinaemic euglycaemic clamp on day 2

SECONDARY OUTCOMES:
change in inflammatory cytokines | Day 1 and 2
  analysis of serum inflammatory markers pre and post procedures on Days 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: David C Wilkinson, FANZCA, Principal Investigator — University of Adelaide
Locations (1):
- Hyperbaric Medicine Unit, Royal Adelaide Hospital, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkinson D, Chapman IM, Heilbronn LK. Hyperbaric oxygen therapy improves peripheral insulin sensitivity in humans. Diabet Med. 2012 Aug;29(8):986-9. doi: 10.1111/j.1464-5491.2012.03587.x. PMID 22269009
- [Background] Wilkinson D, Nolting M, Mahadi MK, Chapman I, Heilbronn L. Hyperbaric oxygen therapy increases insulin sensitivity in overweight men with and without type 2 diabetes. Diving Hyperb Med. 2015 Mar;45(1):30-6. PMID 25964036